CLINICAL TRIAL: NCT00914693
Title: Multicenter, Open-label, Uncontrolled Study to Investigate the Efficacy and Safety of the Transdermal Contraceptive Patch Containing 0.55 mg Ethinyl Estradiol and 2.1 mg Gestodene (Material no. 80876395) in a 21-day Regimen for 13 Cycles in 1650 Healthy Female Subjects
Brief Title: EU/LA Pearl Index Study - Transdermal Contraceptive Patch
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 91554; 2008-004214-27 (EudraCT Number); 310801 (Other: Company internal)
Record Dates: First submitted 2009-05-05; First posted 2009-06-05 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Contraception
Keywords: Fertility control; Contraception
MeSH Terms: interventions — Ethinyl Estradiol; Gestodene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Ethinylestradiol/Gestodene (BAY86-5016)

INTERVENTIONS:
Drug: Ethinylestradiol/Gestodene (BAY86-5016) — 7-day patch containing 0.55 mg ethinylestradiol (EE) and 2.1 mg gestodene (GSD) in a 21-day regimen

SUMMARY:
The aim of the present study is to prove efficacy and safety of a new contraceptive patch.

ELIGIBILITY:
Inclusion Criteria:

* Requiring contraception
* Normal cervical smear
* Smokers not older than 30 years
* History of regular cyclic menstrual periods

Exclusion Criteria:

* Pregnancy or lactation
* Obesity (BMI> 30 kg/m2
* Significant skin reaction to transdermal preparations or sensitivity to surgical / medical tape
* Any disease that may worsen under hormonal treatment (cardiovascular, liver, metabolic)
* Use of other contraceptive methods than study medication

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1694 (Actual)
Dates: Start 2009-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Occurrence of pregnancy | 13 treatment cycles each consisting of 28 days and follow-up period of 14 days

SECONDARY OUTCOMES:
Cervical smear | 13 treatment cycles each consisting of 28 days
Adverse events | 13 treatment cycles each consisting of 28 days
Bleeding pattern and cycle control | 13 treatment cycles each consisting of 28 days

OTHER OUTCOMES:
Treatment compliance | 13 treatment cycles each consisting of 28 days
Subjective assessment of satisfaction with the treatment | 13 treatment cycles each consisting of 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (59):
- Argentina (4):
  - Lanús Oeste, Buenos Aires
  - San Isidro, Buenos Aires
  - Buenos Aires, Ciudad Auton. de Buenos Aires
  - Rosario, Santa Fe Province
- Australia (5):
  - Ashfield, New South Wales
  - Adelaide, South Australia
  - North Adelaide, South Australia
  - Clayton, Victoria
  - Nedlands, Western Australia
- Chile (4):
  - Temuco, Región de la Araucanía
  - Santiago, Santiago Metropolitan
  - Santiago
  - Temuco
- France (7):
  - Biarritz
  - Montargis
  - Nîmes
  - Quetigny
  - Reims
  - Saint-Germain-en-Laye
  - Toulouse
- Germany (13):
  - Frankfurt am Main, Hesse
  - Aachen, North Rhine-Westphalia
  - Cologne, North Rhine-Westphalia
  - Siegen, North Rhine-Westphalia
  - Wuppertal, North Rhine-Westphalia
  - Dippoldiswalde, Saxony
  - Dresden, Saxony
  - Leipzig, Saxony
  - Blankenburg, Saxony-Anhalt
  - Jessen, Saxony-Anhalt
  - Magdeburg, Saxony-Anhalt
  - Berlin, State of Berlin
  - Gera, Thuringia
- Italy (11):
  - Francavilla Fontana, Brindisi
  - Bologna
  - Cagliari
  - Catanzaro
  - Florence
  - Modena
  - Palermo
  - Pavia
  - Perugia
  - Pisa
  - Siena
- Mexico (6):
  - Chihuahua City, Chihuahua
  - Torreón, Coahuila
  - San Luis Potosí City, San Luis Potosí
  - Mexico City
  - México D.F.
  - México, D.F.
- Spain (9):
  - Barcelona, Barcelona
  - San Fernando, Cádiz
  - Lugo, Lugo
  - Pamplona, Pamplona
  - Vigo, Pontevedra
  - Dos Hermanas, Sevilla
  - Alava, Vitoria
  - Zaragoza, Zaragoza
  - Barcelona

REFERENCES:
- See also: Click here and search for Bayer Product information provided by EMA — http://www.clinicaltrialsregister.eu